CLINICAL TRIAL: NCT05504772
Title: Precision Medicine for Every Child With Cancer
Acronym: ZERO2
Status: Recruiting | Type: Observational
Sponsor: Australian & New Zealand Children's Haematology/Oncology Group (Other)
Collaborators: Children's Cancer Institute (CCI) (Unknown); Minderoo Foundation (Unknown); Medical Research Future Fund (Other)
Responsible Party: Sponsor
Other Study IDs: ZERO2
Record Dates: First submitted 2022-01-30; First posted 2022-08-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Childhood Cancer; Childhood Solid Tumor; Childhood Brain Tumor; Childhood Leukemia; Refractory Cancer; Relapsed Cancer
Keywords: children; precision medicine; personalised medicine; molecular profiling; pediatric; paediatric
MeSH Terms: conditions — Neoplasms; Recurrence | interventions — Whole Genome Sequencing; Base Sequence; DNA Methylation; High-Throughput Nucleotide Sequencing; In Vitro Techniques; Liquid Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour, blood, bone marrow, cerebrospinal fluid (CSF), urine, skin biopsy, cytogenetic culture, extracted DNA and peripheral blood stem cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (13):
- High-risk cancers: One of the following two criteria must be met:
  1. Confirmed or suspected high-risk malignancy defined as expected overall survival < 30% based on current literature for the specific cancer
  2. Cancers for which standard therapy would result in unacceptable and severe morbidity (e.g., infantile fibrosarcoma where definitive surgery would require amputation of limb) Note: This does not include HR neuroblastoma at diagnosis as this group of patients have an overall survival ≥30% and belongs to Cohort 4A.
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Genetic: High Throughput Sequencing (in vitro); Genetic: Patient Derived Xenograft (PDX)(in vivo); Other: Liquid Biopsy
- Rare tumors: At least one of the following three criteria must be met:
  1. A rare tumor of uncertain prognosis due to rarity of disease
  2. A rare tumor with no established treatment strategy
  3. A cancer where routine histopathological examination has not been able to establish a diagnosis
  4. Confirmed histiocytic disorder AND molecular profiling may facilitate diagnosis and/or treatment
  5. Confirmed proliferative vascular or lymphatic malformation AND has failed conventional treatment, e.g., surgery or embolization, OR no appropriate treatment is available AND the disease is organ, limb or life threatening, or debilitating
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Primary central nervous system (CNS) tumours: Patient is suspected or confirmed to have a primary CNS tumor, including low and high-grade tumors
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Neuroblastoma: Patient is suspected or confirmed to have neuroblastoma 4A: HR neuroblastoma at diagnosis 4B: Non-HR neuroblastoma
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Acute myeloid leukemia, myelodysplastic syndrome and other leukemias not classified as ALL: Patient is confirmed by flow cytometry to have acute myeloid leukemia (AML) or other leukemias (Note: Verbal confirmation of flow cytometry result is adequate for enrolment)
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Acute lymphoblastic leukemia (ALL): Patient is confirmed to have acute lymphoblastic leukemia by flow cytometry (Note: Verbal confirmation of flow cytometry result is adequate for enrolment)
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Lymphomas: Patient is suspected or confirmed to have a lymphoma
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Sarcomas: Patient is suspected or confirmed to have a sarcoma Includes gastrointestinal stromal tumour (GIST), malignant peripheral nerve sheath tumour (MPNST), desmoplastic small round cell tumour (DSRCT)
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Renal tumors: Patient is suspected or confirmed to have a renal tumor Includes clear cell sarcoma of kidney
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Hepatic and biliary tree tumors: Patient is suspected or confirmed to have a liver or biliary tree tumor
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Thyroid and endocrine tumors: Patient is suspected or confirmed to have a thyroid or endocrine cancer
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Other tumors: Patient is suspected or confirmed to have a tumor which does not fit into any of the above
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy
- Germline only: One of the following two criteria must be met:
  1. Patients whose submitted tumor sample could not yield sufficient DNA for any molecular analysis AND participants/parents have consented to return of germline findings.
  2. Patients who do not have appropriate tumor sample to be submitted for molecular profiling may be considered for germline only analysis. Obtaining tumor samples wherever possible will be encouraged.
  Interventions: Genetic: Whole Genome Sequencing; Genetic: RNA seq; Genetic: DNA Methylation; Genetic: Targeted Panel Sequencing; Other: Liquid Biopsy

INTERVENTIONS:
Genetic: Whole Genome Sequencing — Each tumor sample will be sequenced and analyzed in parallel with its matched normal (germline DNA from the same patient) to enable the identification of somatic aberrations.
Genetic: RNA seq — Results will be used for bioinformatics analysis for fusion transcripts and gene expression.
Genetic: DNA Methylation — Genome-wide assessment of DNA methylation will be conducted on all samples where possible.
Genetic: Targeted Panel Sequencing — Targeted panel sequencing may be performed:
  1. When WGS is not feasible or appropriate, e.g., insufficient DNA from fresh or frozen sample or only Formalin-Fixed Paraffin-Embedded (FFPE) material is available
  2. When mosaicism is suspected
  3. When indicated for a disease type
Genetic: High Throughput Sequencing (in vitro) — High throughput drug screening will be attempted for tumors from Cohort 1 (high-risk cancers with survival <30%) and selected tumor types.
  Groups: High-risk cancers
Genetic: Patient Derived Xenograft (PDX)(in vivo) — In vivo drug testing in patient derived xenograft (PDX) will be attempted for tumors from Cohort 1 (high-risk cancers) and selected tumor types.
  Groups: High-risk cancers
Other: Liquid Biopsy — Liquid biopsy will be investigated as a non-invasive method for diagnosis of tumors that are difficult to biopsy directly, understanding tumor heterogeneity, monitoring of treatment response, and detection of minimal residual disease (MRD)/relapse in leukemia, solid and CNS tumors.

SUMMARY:
To improve outcomes for childhood cancer patients through the implementation of precision medicine.

DETAILED DESCRIPTION:
Through the pilot TARGET and national PRISM trials the feasibility and benefits of using comprehensive molecular profiling and preclinical drug testing in real time for high-risk (HR) patients has been demonstrated. However, the role of precision medicine, especially in facilitating diagnosis and risk stratification in non-HR childhood cancers has not been studied. Integrative tumor-germline whole genome sequencing (WGS) analysis has the potential to advance our understanding of cancer predisposition. In this study, the ZERO platform will be extended to all children with cancer in Australia and New Zealand, evaluating the benefits of precision medicine in different childhood cancer types and risk groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age < 18 years Note: Individual patients aged 19 - 25 years old with a pediatric cancer, e.g., neuroblastoma, may be enrolled after discussion with, and at the discretion of, the Study Chair or their delegate.
2. Life expectancy >6 weeks at time of enrolment
3. Consent i. Signed and dated informed consent for study enrolment from participant aged ≥ 18 years or from parent/guardian of participant aged <18 years. ii. Separate signed and dated informed consent for understanding the role of germline testing and choice for the return of germline results.

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients <18 years of age with a diagnosis of tumor or cancer Patients aged 19 - 25 years with a diagnosis of a pediatric tumor or cancer
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2022-12-16 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Utility of recommended personalized therapy for HR childhood cancer patients. | 5 years
  Disease control rate (stable disease + partial response + complete response) in HR patients who have received recommended personalized therapy which are molecularly and/or preclinically directed
Utility of recommended personalized therapy for non-HR childhood cancer patients. | 5 years
  The proportion of non-HR patients for whom the disease specific, clinically relevant, virtual molecular panel provides additional or equivalent results for diagnosis and risk stratification when compared with routine diagnostic tests.

SECONDARY OUTCOMES:
Utility of pre-defined virtual molecular panel for non-HR childhood cancer patients. | 5 years
  The proportion of non-HR patients for whom a pre-defined virtual molecular panel; leads to a streamline molecular report issued within 4 weeks from receipt of samples, changes or refines the initial histopathological diagnosis, changes or refines risk stratification at diagnosis, changes or refines treatment at diagnosis and/or facilitates enrolment in clinical trials requiring prior molecular studies.
Utility of comprehensive precision medicine for patients with rare tumors in childhood. | 5 years
  Proportion of rare cancer cohort patients for which comprehensive precision medicine improves diagnosis, identifies at least one therapeutic target or facilitates improvement in therapy within a clinically relevant timeframe.
Utility of Molecular Tumour Board (MTB) recommendation tier system for HR childhood cancer patients. | 5 years
  Evaluation of the correlation of MTB recommendation tier to treatment outcome, clinician rated value of MTB recommendation tier in facilitating therapeutic decision and drug access and proportion of HR patients for which the MTB recommendation improves diagnosis, risk stratification or facilitates improvement in therapy within a clinically relevant timeframe.
Utility of preclinical testing in HR childhood cancer patients. | 5 years
  Evaluation of proportion of tumors where in vitro sensitivity testing can be successfully performed compared with PRISM trial, turnaround time for preclinical in vitro and in vivo drug testing, proportion of tumors where in vitro drug sensitivity identifies additional molecular drivers and proportion of patients for whom preclinical testing:
  i. Facilitates therapeutic decision ii. Identifies additional therapeutic options in patients for whom genomic profiling did not identify molecular targets iii. Predicts clinical outcome
Clinical utility of germline WGS in patients with childhood cancers. | 5 years
  Evaluation of;
  1. Proportion of HR and non-HR patients with a reportable germline finding (i. For whom the result was not previously known ii. For whom the results would have been missed using current clinical testing criteria)
  2. Proportion of patients for whom medical management for the current cancer and future cancer risk has been altered based on the germline findings
Treatment outcome in HR childhood cancer patients who have received recommended personalised therapy which are molecularly and/or preclinically directed. | 5 years
  Evaluation of;
  1. Objective response in patients who have received single agent versus combination personalized therapy
  2. Disease control (stable disease + partial response + complete response) in patients who have received a single agent versus combination personalized therapy
  3. Progression-free interval (PFI) ratio: PFI personalized therapy : PFI conventional therapy
  4. Difference in outcome between patients have received recommended personalised therapy and those who did not (i. Proportion of patients without progression or death at 6 and 12 months between the two groups ii. Difference in progression-free and overall survival between the two groups)

CONTACTS AND LOCATIONS:
Overall Officials: David Ziegler, Principal Investigator — SCHN
Locations (11):
- Australia (9):
  - Women's and Children's Hospital, Adelaide
  - Queensland Children's Hospital, Brisbane
  - Royal Hobart Hospital, Hobart
  - Monash Children's Hospital, Melbourne
  - Royal Children's Hospital, Melbourne
  - John Hunter Children's Hospital, Newcastle
  - Perth Children's Hospital, Perth
  - Sydney Children's Hospital, Randwick, Sydney
  - The Children's Hospital at Westmead, Sydney
- New Zealand (2):
  - Starship Children's Hospital, Auckland, Grafton
  - Christchurch Hospital, Christchurch